CLINICAL TRIAL: NCT01584258
Title: International Randomised Study of Prostatectomy vs Stereotactic Body Radiotherapy (SBRT) and Conventionally Fractionated Radiotherapy vs SBRT for Organ-Confined Prostate Cancer
Brief Title: Prostate Advances in Comparative Evidence
Acronym: PACE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: The Institute of Cancer Research, Sutton, Surrey, UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR3766
Record Dates: First submitted 2012-04-22; First posted 2012-04-24 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate adenocarcinoma; Organ-confined prostate cancer; Low-risk prostate cancer; Intermediate-risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Intervention Model Description: Multicentre, international phase 3 randomised controlled study comprising three parallel randomisations with a common experimental arm.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PACE-A: Prostatectomy vs prostate SBRT (Active Comparator): Low and intermediate risk patients, for whom surgery is considered, will be randomised to prostatectomy vs prostate SBRT delivered with 36.25 Gy in 5 fractions.
  Interventions: Procedure: Prostatectomy; Radiation: Prostate SBRT
- PACE-B: Conventionally Fractionated RT vs Prostate SBRT (Active Comparator): Low and intermediate risk patients, for whom surgery is not considered or who refuse surgery, will be randomised to either conventionally fractionated radiotherapy delivered to a dose of 78 Gy in 39 fractions or 62 Gy in 20 fractions vs SBRT delivered with 36.25 Gy in 5 fractions.
  Interventions: Radiation: Conventionally Fractionated Prostate Radiotherapy; Radiation: Prostate SBRT
- PACE-C: Conventionally Fractionated RT vs Prostate SBRT (Active Comparator): Intermediate and high risk patients, indicated for 6 months ADT, will be randomised to either conventionally fractionated radiotherapy delivered to a dose of 60 Gy in 20 fractions vs SBRT delivered with 36.25 Gy in 5 fractions.
  Interventions: Radiation: Conventionally Fractionated Prostate Radiotherapy; Radiation: Prostate SBRT

INTERVENTIONS:
Procedure: Prostatectomy — Radical prostatectomy: performed open, laparoscopically or using a robotically assisted laparoscopic approach.
  Arms: PACE-A: Prostatectomy vs prostate SBRT
Radiation: Conventionally Fractionated Prostate Radiotherapy — Conventional fractionation delivered to a dose of:
  (PACE-B) 78 Gy in 39 fractions or 62 Gy in 20 fractions; (PACE-C) 60 Gy in 20 fractions
  Arms: PACE-B: Conventionally Fractionated RT vs Prostate SBRT; PACE-C: Conventionally Fractionated RT vs Prostate SBRT
Radiation: Prostate SBRT — Prostate SBRT delivered to a dose of 36.25 Gy in 5 fractions.

SUMMARY:
This study is an international multicentre randomised study of low, intermediate, and high risk prostate cancer and is composed of three parallel randomisation schemes based on applicability of surgery as a treatment for the patient and risk group. Low and intermediate risk patients, for whom surgery is a consideration, are randomised to either prostatectomy or prostate SBRT. Low and intermediate risk patients, for whom surgery is not a consideration, are randomised to either conventionally fractionated radiotherapy or prostate SBRT. Intermediate and high risk patients, for whom ADT treatment is indiacted and surgery is not a consideration, are randomised to either conventionally fractionated radiotherapy or prostate SBRT. Efficacy, toxicity and quality of life outcomes will be compared across the pairs in each randomisation.

ELIGIBILITY:
Inclusion critieria (all arms):

* Histological confirmation of prostate adenocarcinoma within the last 18 months (unless on active surveillance and not clinically indicated)
* Men aged ≥18 years at randomisation
* WHO performance status 0 - 2
* Patients considered candidates for surgery are eligible for PACE-A; patients not considered candidates for surgery and patients who decline surgery or prefer to avoid surgery are eligible for PACE-B and PACE-C.
* Ability of the research subject to understand and the willingness to sign a written informed consent document.

Specific risk stratification inclusion criteria for PACE-A and PACE-B:

* Minimum of 10 biopsy cores.
* Gleason score ≤ 3+4
* Clinical and/or MRI stage T1c -T2c, N0-X, M0-X
* PSA ≤ 20 ng/ml (completed within 60 days of randomisation)
* Patients belonging to one of the following risk groups:
* Low risk - patients with tumours meeting all of the following criteria:

  * Gleason ≤ 6
  * Clinical stage T1-T2a
  * PSA < 10 ng/ml (within 60 days prior to randomisation)
* Intermediate risk - patients with tumours meeting any one of the following criteria:

  * Gleason 3+4
  * Clinical stage T2b or T2c
  * PSA 10-20 ng/ml (within 60 days prior to randomisation)

Specific risk stratification inclusion criteria for PACE-C:

* Patient planned for a minimum of 6 months ADT (maximum of 12 months). Patients receiving extended androgen deprivation therapy (18 months maximum) to permit safe delay of radiotherapy as a result of the COVID19 pandemic (only) are eligible.
* Gleason score ≤ 4+4
* MRI stage T1c -T3a, N0-X, M0-X
* PSA ≤ 30 ng/ml (within 60 days prior to starting ADT)
* Patients belonging to one of the following risk groups:
* Intermediate risk - includes the presence of any of the following, assuming no high risk features apply:

  * Gleason 7 (3+4 or 4+3)
  * T2 (N0, M0-X)
  * PSA 10-20 ng/ml
* High risk - patients with tumours that meet a maximum of 2 of the following criteria:

  * Gleason 4+4 (max ≤ 50% cores)
  * T3a (N0, M0)
  * PSA >20 ng/ml

Exclusion criteria (all arms):

* Previous malignancy within the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin), or if previous malignancy is expected to significantly compromise 5 year survival.
* Prior pelvic radiotherapy.
* Prior androgen deprivation therapy (including androgen agonists and antagonists) for PACE-A and PACE-B participants.
* Any prior active treatment for prostate cancer (with the exception of ADT for PACE-C participants). Patients previously on active surveillance are eligible if they continue to meet all other eligibility criteria.
* Life expectancy <5 years.
* Bilateral hip prostheses or any other implants/hardware that would introduce substantial CT artefacts.
* Medical conditions likely to make radiotherapy inadvisable eg inflammatory bowel disease, significant urinary symptoms.
* For patients having fiducials inserted: Anticoagulation with warfarin/ bleeding tendency making fiducial placement or surgery unsafe in the opinion of the clinician.
* Participation in another concurrent treatment protocol for prostate cancer.

Specific exclusion criteria for PACE-C:

* >14 weeks of androgen deprivation therapy prior to randomisation
* Medical conditions likely to make ADT inadvisable (e.g. significant and ongoing cardiac issues).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2205 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PACE-B and PACE-C: Freedom from biochemical or clinical failure | 5 years from randomisation (primary timepoint)
  Biochemical progression is defined as: Phoenix definition
  Clinical progression is defined as: commencement (PACE-B) or re-commencement (PACE-C) of androgen deprivation therapy, local recurrence, nodal recurrence and distant metastases
PACE-A: Co-primary patient reported outcomes of urinary incontinence and bowel bother | 2 years from treatment (primary timepoint)
  Urinary incontinence assessed by the number of absorbent pads required per day to control leakage measured by The Expanded Prostate Cancer Index (EPIC) questionnaire.
  Bowel bother assessed by summary score from the EPIC questionnaire.

SECONDARY OUTCOMES:
All arms: Clinician reported acute toxicity | 10 years
  CTCAE and RTOG (SBRT and conventional RT patients) or Clavien scale (surgical patients).
All arms: Clinician reported late toxicity | 10 years
  CTCAE and RTOG (SBRT and conventional RT patients only).
All arms: Patient reported acute and late bowel, bladder and erectile dysfunction symptoms. | 10 years
  Assessed using International Index of Erectile Function-5 (IIEF-5), International Prostate Symptom Score (IPSS), Vaizey score, and Expanded Prostate Index Composite-26 (EPIC-26) instruments.
All arms: Disease-specific and overall survival | 10 years
  Disease-specific and overall survival
All arms: Progression-free survival | 10 years
  Radiographic, clinical or biochemical evidence of local or distant failure
PACE-A and PACE-B: Commencement of androgen deprivation therapy; PACE-C: Re-commencement of androgen deprivation therapy | 10 years
  LHRH analogues, anti-androgens, orchidectomy
PACE-A: Freedom from biochemical or clinical failure | 5 years from randomisation (primary timepoint)
  Biochemical progression is defined as: Phoenix definition (SBRT arm) or >0.2ng/ml (surgical arm)
  Clinical progression is defined as: commencement of androgen deprivation therapy, local recurrence, nodal recurrence and distant metastases

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas van As, MD, Study Director — Royal Marsden NHS Foundation Trust, London, United Kingdom; Peter Ostler, MD, Principal Investigator — Mount Vernon Cancer Centre, United Kingdom; Alison Tree, MD, Principal Investigator — Royal Marsden NHS Foundation Trust, London, United Kingdom
Locations (68):
- Canada (9):
  - Northeast Cancer Centre, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Walker Family Cancer Centre, Niagara, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Hôpital Charles-LeMoyne, Montreal, Quebec
  - Hôpital Maisonneuve Rosemont, Montreal, Quebec
- Ireland (4):
  - Beacon Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - St. Luke's Hospital, Dublin
- Auckland City Hospital, Auckland, New Zealand
- United Kingdom (54):
  - Hinchingbrooke Hospital, Huntingdon, Cambridgeshire
  - Colchester General Hospital, Colchester, Essex
  - Churchill Hospital, Oxford, Oxfordshire
  - Mount Vernon Cancer Centre, London, Surrey
  - Velindre Cancer Centre, Cardiff, Wales
  - University Hospital Coventry & Warwickshire NHS Trust, Coventry, West Midlands
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Pilgrim Hospital, Boston
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - West Suffolk Hospital, Bury
  - Addenbrooke's Hospital, Cambridge
  - Queen Elizabeth Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - Velindre Hospital, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Royal Derby Hospital, Derby
  - Western General, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - The Beatson, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Ipswich Hospital, Ipswich
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Free Hospital, London
  - Imperial College, London, London
  - Charing Cross Hospital, London
  - Guy's Hospital, London
  - North Middlesex University Hospital, London
  - Royal Marsden NHS Foundation Trust, London
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Maidstone Hospital, Maidstone
  - Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Northampton General Hospital, Northampton
  - Norfolk & Norwich Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Glan Clwyd Hospital, Rhyl
  - Queens Hospital, Romford
  - Weston Park Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - Kings Mill Hospital, Sutton in Ashfield
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Southend University Hospital, Westcliff-on-Sea
  - Worcestershire Royal Hospital, Worcester

REFERENCES:
- [Derived] Tree AC, Hinder V, Chan A, Tolan S, Ostler P, van der Voet H, Kancherla K, Loblaw A, Naismith O, Jain S, Martin A, Price D, Brand D, Chu W, Duffton A, Kelly P, O'Neill B, Staffurth J, Sasso G, Pugh J, Manning G, Brown S, Burnett S, Griffin C, Hall E, van As N; PACE Investigators. Intensity-modulated moderately hypofractionated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-C): early toxicity results from a randomised, open-label, phase 3, non-inferiority trial. Lancet Oncol. 2025 Jul;26(7):936-947. doi: 10.1016/S1470-2045(25)00205-0. Epub 2025 Jun 12. PMID 40517778
- [Derived] Smith RP, Mohammed MA, Beriwal S, Benoit RM. Prostate Brachytherapy With Cs-131: Long-term Results Compared With Published Stereotactic Body Radiotherapy Data. Am J Clin Oncol. 2025 Jan 1;48(1):34-37. doi: 10.1097/COC.0000000000001145. Epub 2024 Oct 17. PMID 39716881
- [Derived] van As N, Griffin C, Tree A, Patel J, Ostler P, van der Voet H, Loblaw A, Chu W, Ford D, Tolan S, Jain S, Camilleri P, Kancherla K, Frew J, Chan A, Naismith O, Armstrong J, Staffurth J, Martin A, Dayes I, Wells P, Price D, Williamson E, Pugh J, Manning G, Brown S, Burnett S, Hall E. Phase 3 Trial of Stereotactic Body Radiotherapy in Localized Prostate Cancer. N Engl J Med. 2024 Oct 17;391(15):1413-1425. doi: 10.1056/NEJMoa2403365. PMID 39413377
- [Derived] Tree AC, Ostler P, van der Voet H, Chu W, Loblaw A, Ford D, Tolan S, Jain S, Martin A, Staffurth J, Armstrong J, Camilleri P, Kancherla K, Frew J, Chan A, Dayes IS, Duffton A, Brand DH, Henderson D, Morrison K, Brown S, Pugh J, Burnett S, Mahmud M, Hinder V, Naismith O, Hall E, van As N; PACE Trial Investigators. Intensity-modulated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-B): 2-year toxicity results from an open-label, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2022 Oct;23(10):1308-1320. doi: 10.1016/S1470-2045(22)00517-4. Epub 2022 Sep 13. PMID 36113498
- [Derived] Brand DH, Tree AC, Ostler P, van der Voet H, Loblaw A, Chu W, Ford D, Tolan S, Jain S, Martin A, Staffurth J, Camilleri P, Kancherla K, Frew J, Chan A, Dayes IS, Henderson D, Brown S, Cruickshank C, Burnett S, Duffton A, Griffin C, Hinder V, Morrison K, Naismith O, Hall E, van As N; PACE Trial Investigators. Intensity-modulated fractionated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-B): acute toxicity findings from an international, randomised, open-label, phase 3, non-inferiority trial. Lancet Oncol. 2019 Nov;20(11):1531-1543. doi: 10.1016/S1470-2045(19)30569-8. Epub 2019 Sep 17. PMID 31540791
- See also: ICR Clinical Trials Unit - PACE website — https://www.icr.ac.uk/our-research/centres-and-collaborations/centres-at-the-icr/clinical-trials-and-statistics-unit/clinical-trials/pace
- See also: Cancer Research UK- PACE — https://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-comparing-surgery-conventional-radiotherapy-and-stereotactic-radiotherapy-for-localised-prostate-cancer-pace